CLINICAL TRIAL: NCT06581770
Title: Evaluation of Validity and Reliability of the Turkish Translation of the Digital Health Readiness Questionaire in Different Chronic Diseases
Status: Recruiting | Type: Observational
Sponsor: Istanbul Galata University (Other)
Collaborators: Biruni University (Other); Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Busra Ulker Eksi, Researcher, Istanbul Galata University
Other Study IDs: AA1234
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Non-Communicable Chronic Diseases; Survey and Questionnaire; Validation Studies; Digital Health
Keywords: digital health; Digital Health Readiness Questionaire
MeSH Terms: conditions — Noncommunicable Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Survey using a questionnaire. — It is a validity and reliability study that can evaluate digital health readiness.
Other: Survey using a questionnaire. — This is a reliability and validity study.

SUMMARY:
The World Health Organization (WHO) defines digital health as the field of knowledge and application related to any aspect of the adoption of digital technology in the stages of improvement. The combination of digital health with technology brings about a new transformation in digital media. This transformation allows for the development of communication and information in health services, the ability to conduct health-related research on digital media and the evaluation of this data. The ease of access to information and the provision of a timely feedback mechanism in the face of problems have enabled the spread of digital health systems, and have also enabled chronic disease management and epidemic disease monitoring.

It is recommended that the term digital readiness be used to cover the combination of digital access and use, digital literacy and digital health literacy. Digital health readiness is also defined as the main determinant of health and is thought to contribute to the improvement of health processes with the development of digital health literacy and to be a useful solution against health problems that may arise in the follow-up of chronic diseases.

Although there are tools in the literature that evaluate digital health readiness, there is no Turkish assessment tool that facilitates the follow-up of non-communicable chronic diseases. Therefore, the aim of our study is to evaluate the translation, validity, and reliability of the Digital Health Readiness Questionaire into Turkish in individuals with chronic non-infectious diseases.

ELIGIBILITY:
Inclusion Criteria:

* The study will include people over the age of 18, native Turkish speakers, literate, obese, diabetic, cardiovascular and respiratory patients.

Exclusion Criteria:

* Individuals with insufficient cooperation (Mini Mental Test score <24) and any cognitive problems that may prevent the administration of the survey will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study aimed to include 200 participants who applied as patients to Istanbul Faculty of Medicine, Department of Internal Medical Sciences, Department of Internal Medicine, Diabetes and Obesity Polyclinic and Istanbul Florence Nightingale Hospital, Department of Cardiovascular Surgery between September 2024 and August 2025 and met the inclusion criteria, based on the ethics committee approvals obtained from Biruni University Clinical Research Ethics Committee, decision number 2015-KAEK-68-22-01 dated 28.07.2022, and the ethics committee approvals obtained from Biruni University Non-Interventional Clinical Research Ethics Committee, decision number 2023/85-65 dated 22.12.2023.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Translation of the digital health readiness questionnaire | 1 month
  Translation of the digital health readiness questionnaire into Turkish and application on the sample

SECONDARY OUTCOMES:
the validity and reliability of the survey in Turkish | 11 months
  To evaluate the translation, validity and reliability of the Digital Health Readiness Survey into Turkish in individuals with chronic non-communicable diseases.

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided